CLINICAL TRIAL: NCT05776654
Title: Characterizing the Recovery Phase of Acute Exacerbations of COPD Using Wearable Remote Monitoring Technology
Brief Title: Wearable Devices in the Recovery Phase of Acute Exacerbations of COPD (AECOPDs)
Status: Completed | Type: Observational
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Responsible Party: Principal Investigator, Bryan Ross, Principal Investigator, McGill University Health Centre/Research Institute of the McGill University Health Centre
Other Study IDs: 2023-8851
Record Dates: First submitted 2023-02-16; First posted 2023-03-20 (Actual); Last update posted 2024-05-29 (Actual); Status verified 2024-05

CONDITIONS: Chronic Obstructive Pulmonary Disease; Chronic Obstructive Pulmonary Disease Exacerbation
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- COPD cohort: Patients with COPD currently experiencing and receiving treatment for an exacerbation.
  Interventions: Device: Biometric wearable devices

INTERVENTIONS:
Device: Biometric wearable devices — Passive data collection using biometric wearable devices.

SUMMARY:
The purpose the study is to successfully characterize the recovery phase of acute exacerbations of COPD in the outpatient setting using remotely captured physiologic data from wearable devices, to compare this with patient self-reported symptom data, to determine which physiologic variable(s) best correspond with AECOPD recovery, and to further document the feasibility, data quantity, data quality, and COPD outpatient usability experience with wearable devices.

ELIGIBILITY:
Inclusion Criteria:

1. Males/females, age ≥40, former/current smokers with ≥10 pack-year smoking history
2. Currently experiencing/receiving treatment for a physician-diagnosed AECOPD
3. Forced expired volume in the first second (FEV1) / Forced vital capacity (FVC) < 0.7 (GOLD 1-4)
4. Ability to provide informed consent

Exclusion Criteria:

1. No existing COPD diagnosis
2. History of cardiac arrhythmia
3. Presence of pacemaker/defibrillator
4. Any medical/cognitive/functional condition which renders inability to don/doff/recharge devices and complete symptom questionnaire
5. Have already received 4 or more days of consecutive corticosteroid and/or antibiotic therapy since presenting to medical attention for their AECOPD

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with COPD currently experiencing an exacerbation.
Sampling Method: Non-Probability Sample
Enrollment: 21 (Actual)
Dates: Start 2023-02-16 (Actual); Primary Completion 2024-01-15 (Actual); Study Completion 2024-01-15 (Actual)

PRIMARY OUTCOMES:
Daily symptom score | Daily for 21 days
  Validated AECOPD symptom score (EXACT PRO) will serve as the dependent (outcome) variable.
Daily/nightly respiration | Daily for 21 days
  Respiratory rate (RR) will serve as the primary independent (predictor) variable, and RR variability will serve as a secondary independent (predictor) variable.

SECONDARY OUTCOMES:
Daily/nightly heart rate and HR variability | Daily for 21 days
  HR and HRV will serve as secondary independent (predictor) variables.
Daily/nightly peripheral body temperature | Daily for 21 days
  Temperature will serve as secondary independent (predictor) variables.
Activity | Daily for 21 days
  Activity parameters (including calories, METS, step count, etc.) will serve as secondary independent (predictor) variables.
Sleep metrics | Daily (nightly) for 21 days.
  Sleep metrics (including rem and non-rem stages of sleep; sleep duration, latency, efficiency, etc.) will serve as secondary independent (predictor) variables.
Autonomic function/Stress | Daily for 21 days
  Metrics of stress/autonomic function (including electrodermal activity) will serve as secondary independent (predictor) variables.

CONTACTS AND LOCATIONS:
Overall Officials: Bryan A. Ross, MD, FRCPC, MSc (Epi, Physiol), Principal Investigator — Research Institute of the McGill University Health Centre (RI-MUHC)
Locations (1):
- McGill University Health Centre, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No
Due to data privacy regulations, individual participant data collected during this study is not publicly accessible. However, access to anonymized data may be granted upon evaluation by the trial management group. Additional documents will also be available upon inquiry. All requests should be directed to the corresponding author (BAR).